CLINICAL TRIAL: NCT06322615
Title: Acupressure for Anxiety: A Pilot Study of a Nurse-Led Acupressure Intervention for Patients Receiving Chemotherapy
Brief Title: Acupressure for Reducing Anxiety in Patients Undergoing Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MC221001; NCI-2024-00538 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 23-004067 (Other: Mayo Clinic Institutional Review Board); MC221001 (Other: Mayo Clinic in Rochester)
Record Dates: First submitted 2024-03-14; First posted 2024-03-21 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Acupressure; Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive Care (acupressure) (Experimental): Patients undergo acupressure over 15-120 seconds at a time for up to 15 minutes. After completion of the session, patients may optionally receive an education session on using acupressure at home.
  Interventions: Procedure: Acupressure Therapy; Other: Educational Intervention; Other: Electronic Health Record Review; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Acupressure Therapy — Undergo acupressure
  Other Names: Acupressure; Ischemic Compression
Other: Educational Intervention — Receive education session about using acupressure at home
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Other: Electronic Health Record Review — Ancillary studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial evaluates whether acupressure is helpful to reduce anxiety related to chemotherapy. Anxiety is experienced by many patients with cancer. Anxiety can be related to chemotherapy and may contribute to other symptoms, such as nausea and poor quality of life. Some patients diagnosed with cancer express interest in non-medicinal ways to manage symptoms. Acupressure is a noninvasive intervention that can be used for many different symptoms. Acupressure is well tolerated with minimal reports of adverse reactions, making it a good choice for patients with cancer. This study may help researchers learn whether acupressure is useful for managing anxiety in patients undergoing chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the feasibility of a nurse- and patient-applied acupressure intervention for patients with anxiety associated with active cancer-directed therapy.

II. Patient-reported changes in acute anxiety associated with both the nurse and self-led acupressure interventions will be ascertained.

OUTLINE:

Patients undergo acupressure over 15-120 seconds at a time for up to 15 minutes. After completion of the session, patients may optionally receive an education session on using acupressure at home.

After completion of study intervention, patients who opted to receive education about using acupressure at home are followed up at 1 week.

ELIGIBILITY:
Inclusion Criteria:

* Be over 18 years of age
* Be actively undergoing chemotherapy in the Mayo Clinic chemotherapy unit
* Report anxiety as a 1 or higher, on a scale from 0 (no anxiety) to 4 (severe anxiety)
* Be willing to undergo a short acupressure session

Exclusion Criteria:

* Does not meet the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-08-08 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Number of patients approached about undergoing acupressure intervention (Feasibility) | Up to 1 year
  Assessed by the number of patients approached about undergoing acupressure intervention.
Number of patients interested in the initial acupressure intervention in the chemotherapy unit (Feasibility) | Up to 1 year
  Assessed by the number of patients who express interest in the initial acupressure intervention in the chemotherapy unit.
Number of patients interested in the home acupressure intervention (Feasibility) | Up to 1 year
  Assessed by the number of patients who express interest in the home acupressure intervention.
Time taken for each nurse-led acupressure intervention in the chemotherapy unit (Feasibility) | Up to 1 year
  Assess by the time recorded for ach nurse-led acupressure intervention in the chemotherapy unit.
Patient-reported changes in acute anxiety | At baseline, after a one-time nurse-administered acupressure session, and after one week of self-administered acupressure sessions
  Assessed with a brief anxiety questionnaire that inquires about the three different domains of anxiety: cognitive symptoms, emotional symptoms, and physical symptoms. Seven questions are answered using 11-point (0-10) scales with different values assigned to the scale per question (e.g. 0=no anxiety/10=worst possible anxiety or 0=strongly disagree/10=strongly agree).

CONTACTS AND LOCATIONS:
Overall Officials: Laura S. Rhee, D.O., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials